CLINICAL TRIAL: NCT00817349
Title: Clinical Registry of the St. Jude Medical Angio-Seal(TM) Evolution(TM) Vascular Closure Device Following Diagnostic and/or Interventional Endovascular Procedures
Brief Title: Angio-Seal Evolution Device Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Vicki Bebeau, Senior Director of Clinical Research, St. Jude Medical
Other Study IDs: 0801
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Vascular Disease; Coronary Artery Disease; Peripheral Artery Disease; Arterial Occlusive Disease; Coronary Heart Disease
Keywords: Angio-Seal; Peripheral vascular disease; Vascular closure device; Arterial closure; Coronary artery disease; Arterial hemostasis; Coronary cardiac catheterization; Percutaneous coronary intervention; Interventional catheterization; Diagnostic catheterization; Common femoral artery; Manual compression; Vascular intervention; Angiogram; Coronary intervention; Coronary angioplasty; Angiography; Arteriotomy; Vascular access
MeSH Terms: conditions — Peripheral Vascular Diseases; Coronary Artery Disease; Peripheral Arterial Disease; Arterial Occlusive Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Collect data on the use of the Angio-Seal Evolution Device in diagnostic and interventional patient populations.

DETAILED DESCRIPTION:
This multi-center clinical registry is designed to collect data on the use of the Angio-Seal Evolution Device in patients who have had diagnostic and/or interventional procedures through femoral artery access. Data will be collected on a patient's initial screening through hospital discharge and 30 days post-procedure to evaluate major and minor vascular complications as defined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient is having a diagnostic and/or interventional procedure via femoral artery access.

Exclusion Criteria:

* Patients who are unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those needing a diagnostic and/or interventional catheterization procedure.
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Collect major vascular complications | 30 days post-procedure

SECONDARY OUTCOMES:
Assess time artery stops bleeding | Immediately following procedure
Collect minor vascular complications | 30 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Robert Applegate, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (10):
- United States (10):
  - Good Samaritan Hospital, Los Angeles, California
  - Michigan Heart, P.C., Ypsilanti, Michigan
  - Cooper Health System, Camden, New Jersey
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Altru Health System Hospital, Grand Forks, North Dakota
  - Ohiohealth Research Institute @ Riverside Methodist Hospital, Columbus, Ohio
  - Providence Health & Services, Portland, Oregon
  - Main Line Health Heart Center: Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Main Line Health Heart Center: Lankenau Hospitals, Wynnewood, Pennsylvania
  - Baptist Hospital West, Knoxville, Tennessee

REFERENCES:
- [Derived] Applegate RJ, Turi Z, Sachdev N, Ahmed A, Szyniszewski A, Foster M, Pratsos A, Shapiro T, Yakubov S, Shavelle D. The Angio-Seal Evolution registry: outcomes of a novel automated Angio-Seal vascular closure device. J Invasive Cardiol. 2010 Sep;22(9):420-6. PMID 20814049